CLINICAL TRIAL: NCT06354608
Title: The Effect of Audio Book and Local Vibration on Pain and Fear in Intramuscular Injection in Children: A Randomised Controlled Study
Brief Title: The Effect of Audio Book and Local Vibration on Pain and Fear in Intramuscular Injection in Children
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Yalova (Other)
Responsible Party: Principal Investigator, Duygu Demir, Assistant Professor, University of Yalova
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: duygudemirr
Record Dates: First submitted 2024-03-12; First posted 2024-04-09 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Procedural Pain
Keywords: Audio Book; Vibration; Intramuscular Injection; pediatric emergency; Child; pain; fear
MeSH Terms: conditions — Pain, Procedural; Pain

STUDY DESIGN:
Intervention Model Description: This study is an experimental, parallel-group (intervention-control), randomized controlled design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Audio Book Group (Experimental): Audiobooks are stories with illustrated stories, and these stories are voiced. Audiobooks are visual and auditory distractions. The researcher will introduce this audio book to both children and parents before the procedure. The child will be allowed to examine the book. Before starting the IM injection procedure, the researcher will show the pages of the book and start the story. The story will be supported by showing the pictures in the book to attract the child's attention. After the child concentrates on the story, the child's leg area where the vastus lateralis muscle is located will be hygienized before the IM injection. During the entire IM injection procedure, the audiobook will continue until the end of the procedure.
  Interventions: Behavioral: Audio Book Group
- Local Vibration Group (Experimental): A local vibration device, an electric vibration device, will be used. During the application, the device must be in full contact with the skin. Local vibration application reduces perceived pain by stimulating nerve fibres according to Melzack and Wall's Gate Control Theory. In the local vibration group, local vibration is applied to the leg area of the child where the vastus lateralis muscle is located for 30 seconds before the IM injection is applied with the vibrating Dolphin massage device. Then, the leg area will be hygienized, and the device will be placed 3-5 cm above the injection area during the procedure, and IM injection will be performed. The device must be in full contact with the skin during the application.
  Interventions: Device: Local Vibration Group
- Control Group (No Intervention): Children in the control group will be received standard care. Control group children will not receive any distraction techniques.

INTERVENTIONS:
Behavioral: Audio Book Group — Audiobook will be applied during the entire IM injection procedure and until the end of the procedure. After the procedure is over, the children will be taken to the waiting area. After being allowed to rest for 1-2 minutes, the child will be asked to rate their level of pain and fear during the procedure. A parent who is with the child and observes the child's behavior, and the same nurse who is independent from the study, will independently rate the child's pain and fear level during the procedure.
  Arms: Audio Book Group
Device: Local Vibration Group — In the local vibration group, IM injection will be performed with a vibrating massage device. After the procedure is finished, the children will be taken to the waiting section. After being allowed to rest for 1-2 minutes, the child will be asked to rate their level of pain and fear during the procedure. A parent who is with the child and observes the child's behavior and the same nurse who is independent from the study will independently rate the pain and fear level of the child during the procedure.
  Arms: Local Vibration Group

SUMMARY:
The study is conducted based on a randomized controlled experimental design to determine the effect of an audio book and local vibration on intramuscular injection in pediatric emergency unit patients aged 4-6 years on pain and fear.

DETAILED DESCRIPTION:
IM injection is one of the medical procedures that causes pain and fear in children. It has been reported that the effect of children's previous pain and fearful experiences continues into adulthood, and this may lead to the avoidance of subsequent medical procedures as a reaction to increased pain and fear. For all these reasons, pediatric nurses and other healthcare professionals should aim for successful pain control before and during painful procedures in children to prevent future adverse effects of painful medical procedures.

Reducing the emotional impact of painful procedures in clinical practice through better pain control is very important for children. Therefore, all healthcare professionals, especially nurses, as the first person to welcome children into the hospital and the person who spends the most time with the child, have important responsibilities in eliminating children's fear of medical procedures. It is very important for pediatric nurses to use nonpharmacological techniques to reduce pain in the IM injection procedure. It is known that non-pharmacological pain control methods help the child cope with pain, reduce pain, and alleviate distress from invasive procedures. The most commonly used of these approaches is the distraction technique, also known as the distraction technique, which is constructed with cognitive and behavioral processes. These include relaxation techniques, deep breathing, listening to music, singing and talking, watching cartoons, games, vibration and cold applications, and distraction cards. As understood from the studies, nonpharmacological approaches help the child cope with the pain experienced in invasive interventions and provide less pain.

It is critical that all pediatric nurses and other healthcare workers who work with children learn about and practice pain-reduction techniques. When the literature was reviewed, it was discovered that there were no studies comparing audiobook and local vibration application to reduce pain and fear perceived during IM injections administered to pediatric patients, whereas there were a limited number of studies evaluating the methods independently. It is thought that there is a need for planning randomized controlled experimental nursing studies in this field. This study is planned to determine the effect of the use of audio book and local vibration on the pain and fear experienced by children during intramuscular injection in children aged 4-6 years. While the population of the study consisted of pediatric patients aged 4-6 years in the pediatric emergency unit between October 2023 and April 2024, the sample consisted of 120 children who met the sample selection criteria. The research consists of 3 groups. These groups will audio book group (n=40), local vibration group (n=40), and control group (n=40). In order for the groups to be distributed homogeneously, the order produced by a computer program (http://www.randomization.com, Balanced permutation) was used. Patients who meet the inclusion criteria and agree to participate in the study assigned to the experimental and control groups according the randomization list. The control variable of the study is demographic characteristics of the children. The dependent variables of the study are pain and fear score. The data are collected using Introductory Information Form, Wong-Baker FACES Pain Scale (W-BPS), Children's Fear Scale (CFS).

ELIGIBILITY:
Inclusion Criteria:

* The child and family agree to participate in the research,
* The child is between the ages of 4-6,
* The child does not have a chronic and mental health problem,
* Absence of visual, auditory problems or mental retardation at a level that can fill the scales,
* No history of sedative, analgesic or narcotic substance use within 24 hours before admission,
* Absence of a disease causing chronic pain,
* Not having a febrile illness at the time of application,
* Being treated in the pediatric emergency unıt at the time of the study,
* Intramuscular injection in the vastus lateralis region,
* Ondansetron will be injected intramuscularly in the vastus lateralis area, as directed by the doctor.
* Performing the operation at once.

Exclusion Criteria:

* The child and family's refusal to participate in the research,
* Having a visual and auditory problem
* The child is less than 4 years old or older than 6 years old
* The child has a chronic and mental health problem
* The child experiences pain,
* To have taken analgesic medication in the last 6 hours.

Ages: 4 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-06-21 (Actual); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
Comparison of the pain score values of the groups Pain assesed by Wong-Baker FACES | Pain levels of the children will be evaluated 1 minute after the procedure.
  The Wong-Baker Faces Pain Scale revised (W-BFS) is used to determine the level of pain during the procedure. The W-BFS is a scale that is most commonly used in identifying pain in children of the ages 3 to 18. It is reported that the scale is reliable when used with children older than the age of 3 who can verbally express the degree of pain they feel. The scale is made up of faces and numbers. Pain is assessed on a scale of "0" to "10." Pain is described by selecting the facial expression depicting the degree of perceived pain. This scale will be assessed independently by the child, a parent who is present and observes the child's behavior, and the same nurse who is independent of the study.
Comparison of the fear score values of the groups | Children's fear levels will be evaluated first 1 minutes before the procedure.
  The Children's Fear Scale (CFS) is used to measure the child's fear level. This scale is a one-item self-report measure for measuring pain-related fear in children. The CFS is a scale from 0 to 4, showing 5 facial expressions ranging from a neutral expression (0 = no anxiety) to a frightened face (4=severe anxiety). CFS is administered by the researcher to the children to assess their fear levels before and after the IM procedure.
Comparison of the fear score values of the groups | Children's fear levels will be evaluated 1 minutes after the procedure.
  The Children's Fear Scale (CFS) is used to measure the child's fear level. This scale is a one-item self-report measure for measuring pain-related fear in children. The CFS is a scale from 0 to 4, showing 5 facial expressions ranging from a neutral expression (0 = no anxiety) to a frightened face (4=severe anxiety). CFS is administered by the researcher to the children to assess their fear levels before and after the IM procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Duygu Demir, Assis. Prof., Study Director — Director; Derya Kılıç, Assis. Prof., Principal Investigator — Researcher
Locations (1):
- University of Yalova, Yalova, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McMurtry CM, Noel M, Chambers CT, McGrath PJ. Children's fear during procedural pain: preliminary investigation of the Children's Fear Scale. Health Psychol. 2011 Nov;30(6):780-8. doi: 10.1037/a0024817. Epub 2011 Aug 1. PMID 21806301
- [Result] Gerceker GO, Binay S, Bilsin E, Kahraman A, Yilmaz HB. Effects of Virtual Reality and External Cold and Vibration on Pain in 7- to 12-Year-Old Children During Phlebotomy: A Randomized Controlled Trial. J Perianesth Nurs. 2018 Dec;33(6):981-989. doi: 10.1016/j.jopan.2017.12.010. Epub 2018 Mar 17. PMID 29559294
- [Result] Ozalp Gerceker G, Ayar D, Ozdemir EZ, Bektas M. Effects of virtual reality on pain, fear and anxiety during blood draw in children aged 5-12 years old: A randomised controlled study. J Clin Nurs. 2020 Apr;29(7-8):1151-1161. doi: 10.1111/jocn.15173. Epub 2020 Jan 22. PMID 31889358
- [Result] Sivri Bilgen B, Balci S. The Effect on Pain of Buzzy(R) and ShotBlocker(R) during the Administration of Intramuscular Injections to Children: A Randomized Controlled Trial. J Korean Acad Nurs. 2019 Aug;49(4):486-494. doi: 10.4040/jkan.2019.49.4.486. PMID 31477677
- [Result] Sunitha Suresh BS, De Oliveira GS Jr, Suresh S. The effect of audio therapy to treat postoperative pain in children undergoing major surgery: a randomized controlled trial. Pediatr Surg Int. 2015 Feb;31(2):197-201. doi: 10.1007/s00383-014-3649-9. Epub 2015 Jan 3. PMID 25555856